CLINICAL TRIAL: NCT03561155
Title: Effects of High-intensity Robot-assisted Training in Hand Function Recovery and ADL Independence in Individuals With Multiple Sclerosis: a Randomized Controlled Single-blinded Trial
Brief Title: Robot-assisted Arm Training in Multiple Sclerosis
Acronym: RAMSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Professor, Universita di Verona
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FISM 14/14/F14
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis; Rehabilitation
Keywords: Upper Extremity; Recovery
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot assisted treatment (Experimental): The experimental group (EG) will undergo a robot-assisted arm training using Amadeo® (Tyromotion-Austria).
  Interventions: Device: Robot assisted treatment (Amadeo®)
- Conventional treatment (Active Comparator): The conventional group (CG) will undergo robot unassisted treatment (Conventional treatment).
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Robot assisted treatment (Amadeo®) — The protocol will consist of exercises as follows:
  passive modality , passive/plus modality , assisted therapy and Balloon.
  Other Names: Robot assisted treatment
  Arms: Robot assisted treatment
Other: Conventional treatment — The protocol will consist of exercises as follow:
  upper limb mobilization, facilitation of movements and active tasks. The exercises will be focused on improving muscle strength, finger extension and flexion and motor control
  Arms: Conventional treatment

SUMMARY:
The upper limb (UL) plays an important role in the daily functioning of patients with Multiple Sclerosis (MS) and negatively influences their quality of life. Effective arm-hand training programs are needed. Various robotic systems have been developed for UL rehabilitation, mainly used in patients with stroke. Preliminary work in MS has focused on proximal sections of the arm. No study has evaluated the use of robotics for improving manual dexterity and their effects on cortical activity. The results of this research project could be relevant for the advancement of knowledge about UL functional recovery in individuals with MS and to determine the pattern of muscle activation underlying functional recovery.

DETAILED DESCRIPTION:
Studies regarding the effectiveness of conventional and robot-based upper limb (UL) rehabilitation in individuals with MS is very limited.In the last 15 years, conventional rehabilitation of the UL in patients with neurological disorders has been enriched by the development of robots as they can provide high-intensity, repetitive, interactive and task-specific exercises.They are increasingly used in rehabilitation after stroke, therefore may also be good candidates for neuromotor rehabilitation of patients with MS. Furthermore, these devices can provide various feedbacks that can guide patients during the sensorimotor training and allow quantitative measurement of motor performance during training.One of these devices is the Amadeo®, a modern, mechatronic end-effector robotic device designed to improve sensorimotor functions in patients with restricted movement in individual fingers or in the entire hand.Another important issue concerns cortical plasticity, which plays a fundamental role in motor learning and neurorehabilitation.To date, the specific mechanisms leading to UL recovery after neurological rehabilitation are still unclear.The development of new EEG instruments allows brain activity to be tested under specific rehabilitation tasks contributes to give new insight in the dynamics of cortical networks reorganization promoted by rehabilitation.The main aim of the study is to perform a single blind RCT on 60 outpatients with MS (age:18-65 years;EDSS<8) in order to compare the efficacy of high-intensity robot-assisted training with conventional treatment on sensorimotor hand recovery, disability in ADLs and QoL.The secondary aim is to explore the underlying neuronal mechanisms of UL recovery by using EEG investigations and innovative robotic equipment. 10 controls (age 18-65 yrs) will undergo one session of the same Video-EEG acquisition to collect normative data to compare with data collected on patients.Each participant will receive 40-minute sessions over an 8 week period (3 days/week). Each session will consist of 30 minutes of hand training and 10 minutes of passive upper limbs mobilization.The experimental group will receive robot-assisted therapy by Amadeo.The control group will receive conventional rehabilitation.Before treatment, immediately after treatment, 1 month after treatment patients will be evaluated with a comprehensive protocol of all ICF domains as well as acquisition by Video-EEG acquisition combined with Amadeo® robotic training device.Primary outcome measures:Fugl-Meyer Assessment Motor Scale.Secondary measures: UL electromyographic analysis,Tremor Severity Scale, Nine Hole Peg Test, Amadeo® hand muscle strength (Newton), Motricity Index, Visual anolgue Scale for tiredness and fatigue; TEMPA, Motor Activity Log, Action Research Arm test, Multiple Sclerosis Quality of Life-54 and the assessment of Life Habits. Parametric tests and nonparametric tests will be performed according to variable distribution (p<.05)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* EDSS score<8
* Mini Mental State Evaluation (MMSE) score>24
* Ashworth Scale Score<2 evaluated at the elbow, wrist and fingers
* Nine Hole Peg Test (NHPT) score >30 sec.

Exclusion Criteria:

* Disease recurrence that worsened significantly during the 3 months prior to recruitment
* Medical therapy not well defined
* Musculoskeletal impairments or excessive pain in any joint that could limit participation in an exercise program
* Severe visual dysfunction
* Performance of any type of rehabilitation treatment in the month prior to recruitment
* Other concomitant neurological or orthopaedic diseases involving the UL and interfering with their function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Action Research Arm test | Up to 6 weeks
  Assesses upper limb functioning using observational methods

SECONDARY OUTCOMES:
Fugl-Meyer Assessment Motor Scale - Arm Section | Up to 6 weeks
  Evaluates and measures recovery in post-stroke hemiplegic patients
Motor Activity Log | Up to 6 weeks
  Semi-structured interview to assess arm function.
Tremor Severity Scale | Up to 6 weeks
  A clinical rating scale which measured the severity of tremor
Nine Hole Peg Test | Up to 6 weeks
  Measures finger dexterity
Motricity Index | Up to 6 weeks
  Measures of strength in upper limb
Amadeo® hand muscle strength (Newton) | Up to 6 weeks
  Measures of muscle strenght using the robotic device
Visual anolgue Scale for tiredness and fatigue | Up to 6 weeks
  Measures of tirediness and fatigue on a 10-point likert scale
Multiple Sclerosis Quality of Life-54 | Up to 6 weeks
  Measures of a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument.
Assessment of Life Habits | Up to 6 weeks
  Assesses participants on 77 life habits from daily activities to social participation across 12 domains.
UL electromyographic analysis of muscle activation | Up to 6 weeks
  Instrumental assessment of muscle activity during a reaching task

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, Professor, Principal Investigator — Universita di Verona
Locations (1):
- UOC Neurorehabilitation, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gandolfi M, Vale N, Dimitrova EK, Mazzoleni S, Battini E, Benedetti MD, Gajofatto A, Ferraro F, Castelli M, Camin M, Filippetti M, De Paoli C, Chemello E, Picelli A, Corradi J, Waldner A, Saltuari L, Smania N. Effects of High-intensity Robot-assisted Hand Training on Upper Limb Recovery and Muscle Activity in Individuals With Multiple Sclerosis: A Randomized, Controlled, Single-Blinded Trial. Front Neurol. 2018 Oct 24;9:905. doi: 10.3389/fneur.2018.00905. eCollection 2018. PMID 30405526